CLINICAL TRIAL: NCT06948786
Title: PROMOTE-FL: Pirtobrutinib and Mosunetuzumab to Enhance Treatment Efficacy for Patients With Relapsed/Refractory Follicular Lymphoma
Brief Title: Pirtobrutinib and Mosunetuzumab for the Treatment of Relapsed/Refractory Grades 1-3A Follicular Lymphoma, PROMOTE-FL Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125134; NCI-2025-02708 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20877 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3a Follicular Lymphoma; Recurrent Follicular Lymphoma; Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — pirtobrutinib; Biopsy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pirtobrutinib, mosunetuzumab) (Experimental): Patients receive pirtobrutinib PO QD on 7 days prior to the start of mosunetuzumab (day -7) and continue it until up to 52 weeks. Patients receive mosunetuzumab intravenously (IV) on days 1, 8, and 15 of cycle 1 then on day 1 of remaining cycles. Cycles of mosunetuzumab repeat every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients with a CR after cycle 8 discontinue mosunetuzumab. Patients also undergo blood sample and oral swab and/or rectal swab collection, tissue biopsy, CT, and PET/CT throughout the study. Additionally, patients may undergo bone marrow aspiration and biopsy at screening and after cycle 8.
  Interventions: Drug: Pirtobrutinib; Biological: Mosunetuzumab; Procedure: Biospecimen Collection; Procedure: Biopsy Procedure; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Pirtobrutinib — Given PO
  Other Names: BTK Inhibitor LOXO-305; LOXO 305; Jaypirca; LY3527727
Biological: Mosunetuzumab — Given IV
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody BTCT4465A; BTCT-4465A; CD20/CD3 BiMAb BTCT4465A; Lunsumio; RG 7828; RG-7828
Procedure: Biospecimen Collection — Undergo blood sample and oral swab and/or rectal swab collection
  Other Names: Biological Sample Collection
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Bx
Procedure: Computed Tomography — Undergo CT and PET/CT
  Other Names: CT Scan; CT; CAT Scan
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: PET scan; PET
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well pirtobrutinib and mosunetuzumab work in treating patients with grade 1-3a follicular lymphoma (FL) that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Pirtobrutinib, a type of tyrosine kinase inhibitor, works by blocking the action of the Bruton tyrosine kinase (BTK) protein. The BTK protein signals cancer cells to multiply, and blocking it may help keep cancer cells from growing. It could also improve T cell fitness and decrease inflammation, therefore, may improve the efficacy and safety of T cell-based therapies, such as mosunetuzumab. Mosunetuzumab is a bispecific antibody that binds both T cells and the lymphoma cancer cells and harnesses T cells to interfere with the ability of cancer cells to grow and spread. Giving pirtobrutinib and mosunetuzumab together may kill more tumor cells in patients with relapsed or refractory grade 1-3a FL and potentially decreases some side effects of mosunetuzumab which are related to T cells being activated (e.g., cytokine release syndrome).

DETAILED DESCRIPTION:
OUTLINE:

Patients receive pirtobrutinib orally (PO) once daily (QD) on 7 days prior to the start of mosunetuzumab (day -7) and continue it until up to 52 weeks. Patients receive mosunetuzumab intravenously (IV) on days 1, 8, and 15 of cycle 1 then on day 1 of remaining cycles. Cycles of mosunetuzumab repeat every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients with a CR after cycle 8 discontinue mosunetuzumab. Patients also undergo blood sample and oral swab and/or rectal swab collection, tissue biopsy (optional), computed tomography (CT), and positron emission tomography (PET)/CT throughout the study. Additionally, patients may undergo bone marrow aspiration and biopsy at screening and after cycle 8.

After completion of study treatment, patients are followed up at 30 days then at standard of care intervals for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand, willing, and capable of signing a written informed consent document
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically confirmed FL, grades 1-3a
* Relapsed after or failed to respond to at least two prior lines of systemic therapy and had received prior treatment with an anti-CD20-directed therapy
* Prior treatment-related adverse events (AEs) must have recovered to grade ≤ 1 with the exception of alopecia and grade 2 peripheral neuropathy
* At least one bi-dimensionally measurable lesion (≥ 1.5 cm in its largest dimension for nodal lesions, or ≥ 1.0 cm in its largest dimension for extranodal lesions within 6 weeks of screening by PET/CT scans with diagnostic computed tomography [CT] scan. PET/magnetic resonance imaging [MRI] scans may be allowed only if they are approved by the principal investigator [PI])
* Aspartate aminotransferase and alanine aminotransferase ≤ 3 x the upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 x ULN; or total bilirubin ≤ 3 x ULN in patients with documented liver involvement or in patients with a documented history of Gilbert syndrome
* Platelet count ≥ 75 000/mm^3 without transfusion within 14 days prior to first dose of pirtobrutinib
* Absolute neutrophil count ≥ 1000/mm^3 in the absence of growth factor support
* Total hemoglobin ≥ 10 g/dL without transfusion within 21 days prior to first dose of pirtobrutinib
* Patients who did not meet criteria for hematologic function because of extensive marrow involvement of non-Hodgkin lymphoma, splenic sequestration, and/or disease-related cytopenia (e.g., immune thrombocytopenia) could be enrolled into the study if they have platelet count ≥ 50,000/mm^3, absolute neutrophil count ≥ 750/mm^3, and hemoglobin ≥ 7.5 g/dL after discussion with and confirmation by the PI
* Activated partial thromboplastin time (or partial thromboplastin time) and prothrombin (or international normalized ratio) ≤ 1.5 ULN
* Estimated creatinine clearance (CL) ≥ 30 mL/min by Cockcroft-Gault formula: (140 - age) x body weight (kg) x 0.85 (if female) serum creatinine (mg/dl) x 72 or other institutional standard methods (e.g., based on nuclear medicine renal scan)
* Negative serum pregnancy test within 3 days of initiating pirto for women of childbearing potential (WOCBP), defined as following: menarche and who are not postmenopausal (and 2 years of non-therapy-induced amenorrhea) or surgically sterile
* Fertile male and WOCBP patients must be willing to use highly effective contraceptive methods from the initiation of study treatment, until at least 3 months after the last dose of mosun or at least one month after the last dose of pirto, whichever occurs last

Exclusion Criteria:

* Prior BTK inhibitor (BTKi) refractory disease defined as disease progression or recurrence during or within 6 months of prior BTKi therapy. If disease progression or recurrence occurs > 6 months after patients are off BTKi (e.g., due to intolerance), it is not considered as BTKi refractoriness. Patients with prior BTKi exposure but not meeting the criteria of BTKi refractoriness can be enrolled in this trial
* Prior exposure to pirtobrutinib
* CD3 T-cell engager exposed disease. However, these patients may be eligible if they stay in remission for at least 24 months after the last treatment with CD3 T-cell engager and have histologically confirmed CD20 expression on lymphoma at relapse or progression of disease
* Prior use of any monoclonal antibody, radioimmunoconjugate or antibody-drug conjugate within 4 weeks before first pirtobrutinib administration
* Prior treatment with systemic immunotherapeutic agents for which the mechanism of action involves T cells, including but not limited to cytokine therapy and anti-CTLA-4, anti-programmed death (PD)-1 and anti-PD-ligand 1 therapeutic antibodies, within 12 weeks or 5 half-lives of the drug, whichever was shorter, before first pirtobrutinib administration
* Treatment with any chemotherapeutic agent, or treatment with any other anti-cancer agent (investigational or otherwise) within 4 weeks or 5 half-lives of the drug, whichever was shorter, prior to first pirtobrutinib administration
* Treatment with radiotherapy within 2 weeks prior to the first pirtobrutinib administration. If patients received radiotherapy within 4 weeks prior to the first pirtobrutinib administration, patients must have had at least one measurable lesion outside of the radiation field. Patients who had only one measurable lesion that was previously irradiated but subsequently progressed are eligible
* History of allogeneic or autologous stem cell transplant (SCT) or chimeric antigen receptor-modified T cell (CAR-T) therapy within 60 days of enrollment or presence of any of the following, regardless of prior SCT and/or CAR-T therapy timing:

  * Active graft versus host disease (GVHD);
  * Cytopenia from incomplete blood cell count recovery post-transplant;
  * Need for anti-cytokine therapy for toxicity from CAR-T therapy; residual symptoms of neurotoxicity > grade 1 from CAR-T therapy;
  * Ongoing immunosuppressive therapy (> 20 mg prednisone or equivalent daily) or have been off immunosuppressive agents < 2 months
* Prior solid organ transplantation
* Patients who cannot swallow oral medications
* History of bleeding diathesis
* Patients who experienced a major bleeding event on prior treatment with a BTKi
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the study drug
* History of autoimmune disease, including but not limited to myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
* Patients with history of macrophage activation syndrome/hemophagocytic lymphohistiocytosis (HLH)
* Patients with history of confirmed progressive multifocal leukoencephalopathy
* History of severe allergic or anaphylactic reactions to monoclonal antibody or BTKi therapy
* History of other malignancy except for the following: history of second malignancy unless in remission for at least 2 years; in-situ carcinomas not requiring treatment intervention, non-melanoma skin cancer curatively treated, nonmetastatic breast, or nonmetastatic prostate cancer where hormonal therapy is being continued as standard of care are allowed
* Current or past history of central nervous system (CNS) lymphoma
* Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease. Patients with a history of stroke who had not experienced a stroke or transient ischemic attack in the past 2 years and had no residual neurologic deficits as judged by the investigator were allowed. Patients with a history of epilepsy who had no seizures in the past 2 years while not receiving any anti- epileptic medications were allowed in the expansion cohorts only
* Significant cardiovascular disease defined as:

  * Unstable angina or acute coronary syndrome within the past 2 months prior to enrollment;
  * History of myocardial infarction within 3 months prior to enrollment;
  * Documented left ventricular ejection fraction (LVEF) by any method of ≤ 40% in the 12 months prior to enrollment;
  * ≥ grade 3 New York Heart Association (NYHA) functional classification system of heart failure;
  * Uncontrolled or symptomatic arrhythmias
* Significant active pulmonary disease (eg, bronchospasm and/or obstructive pulmonary disease)
* Known active and uncontrolled bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to first pirtobrutinib administration
* Known or suspected chronic active Epstein Barr virus infection
* Known active cytomegalovirus (CMV) infection. Unknown or negative status are eligible
* Recent major surgery within 4 weeks prior to first pirtobrutinib administration
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection based on criteria below:

  * Hepatitis B virus (HBV):

    * Patients with positive hepatitis B surface antigen (HBsAg) are excluded
    * Patients with positive hepatitis B core antibody (anti-HBc) and negative HBsAg require a negative hepatitis B polymerase chain reaction (PCR) evaluation before enrollment
    * Patients who are HBV deoxyribonucleic acid (DNA) PCR positive will be excluded
  * Hepatitis C virus (HCV): If positive hepatitis C antibody result, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA) before enrollment. Patients who are hepatitis C RNA positive will be excluded
* Patients who have tested positive for human immunodeficiency virus (HIV) are excluded due to risk of opportunistic infections with both HIV and BTK inhibitors. For patients with unknown HIV status, HIV testing will be performed at Screening and result must be negative for enrollment
* Patients requiring therapeutic anticoagulation with warfarin or another vitamin K antagonist
* Pregnant or breast-feeding women
* Administration of live vaccination within 28 days of first administration of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2031-07-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) rate | After cycle 8 of mosunetuzumab (cycle length = 21 days)
  Will report the number of CR and the estimated CR rate with 95% exact binomial confidence interval (CI). Will build logistic regression to evaluate the risk factor association with the endpoint of interest.
Progression free survival (PFS) | From trial enrollment to disease progression or death, whichever occurs first, assessed at 1 year
  Analyses will follow standard methodology by employing Kaplan-Meier (KM) and Cox proportional hazard model methodology. The 1-year PFS rate and 95% CI will be estimated by KM.

SECONDARY OUTCOMES:
Cytokine release syndrome (CRS) | Up to 30 days after last dose of study treatment
  CRS will be graded by the American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading system. The rate and grade of CRS will be reported.
Immune effector cell-associated neurotoxicity syndrome (ICANS) | Up to 30 days after last dose of study treatment
  ICANS will be graded by the ASTCT Consensus Grading system. Will report the rate and grade of ICANS.
Incidence of grade 3 or higher adverse events (AEs) | Up to 30 days after last dose of study treatment.
  AEs will be graded in severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Overall survival | From trial enrollment to death from any cause, assessed up to 4 years
  Analyses will follow standard methodology by employing KM and Cox proportional hazard model methodology.
Event free survival | From trial enrollment to death from any cause, disease progression, needing the next line of therapy, whichever occurs first, assessed up to 4 years
  Analyses will follow standard methodology by employing KM and Cox proportional hazard model methodology.
Overall response | After 8 cycles of mosunetuzumab (cycle length = 21 days)
  Will report the count and percentage with 95% CI of patients who achieve overall response, including CR and partial response (PR).
Duration of response | From first PR or CR to progression of disease or death, whichever occurs first, assessed up to 4 years
  Analyses will follow standard methodology by employing KM and Cox proportional hazard model methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Mengyang Di, MD, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No